CLINICAL TRIAL: NCT01988168
Title: Closure of Skin in ChorioAmnionitis Research Pilot Study
Acronym: CSCAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Ellen Giesbrecht, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-03009
Record Dates: First submitted 2013-10-31; First posted 2013-11-20 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Chorioamnionitis; Pregnancy Complications, Infectious; Complications; Cesarean Section; Postoperative Complications
Keywords: Suture Techniques; Sutures; Surgical Staplers
MeSH Terms: conditions — Chorioamnionitis; Pregnancy Complications, Infectious; Postoperative Complications | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suture closure (Experimental): Closure of skin with a running subcuticular, absorbable monofilament suture.
  Interventions: Procedure: Suture closure
- Staples closure (Active Comparator): Closure of skin with stainless-steel surgical staples.
  Interventions: Procedure: Staples closure

INTERVENTIONS:
Procedure: Suture closure — A running subcuticular suture is placed by taking horizontal bites through the papillary dermis on alternating sides of the wound. An absorbable suture is used and left in place until degraded and absorbed by the patient's tissues.
  Other Names: 3-0 Monocryl suture (from Ethicon)
  Arms: Suture closure
Procedure: Staples closure — Surgical stapling devices re-appose skin edges with stainless steel or titanium staples. A second operator everts the wound skin edges while the operator applies staples along the incision. Staples can be removed on post-operative day 2 or 3, or delayed further according the surgeon preference based on patient characteristics.
  Arms: Staples closure

SUMMARY:
The purpose of the CSCAR pilot study is to improve the design of a full-scale trial by determining the patient recruitment rate and participation rate. The objective of the full-scale trial is to determine the optimal method of skin closure after Caesarean delivery in women with chorioamnionitis, which is an acute inflammation of the membranes and chorion of the placenta, seen typically after rupture of membranes with ascending polymicrobial bacterial infection. Women in labour with chorioamnionitis will be randomized at the time of Caesarean delivery to skin closure with either staples or sutures. The women will be followed at 6 weeks and 6 months post-partum in order to establish the occurrence of surgical site infection and wound disruption, as well as evaluation of the scar and other secondary questions.

The investigators hypothesis is that closure of skin with sutures will have a rate of wound infection that is no higher than the rate of wound infection when closing skin with staples. The investigators also hypothesize that closure with sutures will have a decreased rate of wound disruption, increased patient satisfaction and decreased length of hospital stay compared to skin closure with staples.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chorioamnionitis (Fever ≥ 38.0°C AND at least TWO of: Maternal tachycardia: Heart rate > 100bpm, Fetal tachycardia: Baseline heart rate > 160bpm, Uterine tenderness, Foul smelling / purulent vaginal discharge, White Blood Cell count > 15,000 cells/mm3)
* Caesarean delivery with Pfannenstiel incision
* Pregnancies >24 weeks
* Scheduled or non-elective procedures
* Primary or repeat Caesarean delivery
* No restrictions based on BMI
* No exclusions due to DM (GDM or non GDM)
* No exclusions due to multiple gestation pregnancy

Exclusion Criteria:

* Non-Pfannenstiel incision
* Immune compromising disease
* History of keloid formation
* Chronic steroid use
* Allergy to staples
* Planned postpartum care at another facility

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient recruitment rate | 1 year
  The patient recruitment rate will be calculated as the total number of women successfully recruited to the trial divided by the total duration of the trial.

SECONDARY OUTCOMES:
Follow-up rates | 6 months post-operative
  Number of women successfully contacted at 6 weeks and at 6 months post-partum divided by the total number of women randomized in the trial
Wound infection | 6 months post-operative
  Number of women who experience a wound infection divided by the total number of eligible women who participate in the trial.
Wound disruption | 6 months post-operative
  Number of women who experience a wound disruption divided by the total number of eligible women who participate in the trial.
Wound cosmesis | 6 months post-operative
  Wound cosmesis will be assessed using the POSAS Observer scale, which is directed at physicians, and the POSAS Patient scale, which is directed at patients
Patient satisfaction | 6 months post-operative
  Using the POSAS Patient Scale, patient satisfaction will be assessed.
Participation rate | 1 year
  The trial participation rate will be calculated as the percentage of eligible women who agreed to participate in the trial divided by the total number of eligible women approached to participate in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Giesbrecht, MD, Principal Investigator — Clinical Assistant Professor, Division of General Gynaecology & Obstetrics, Department of Obstetrics and Gynaecology, University of British Columbia; Site Head, Department of Obstetrics, BC Women's Hospital; Jennifer A Hutcheon, PhD, Study Director — Assistant Professor, Division of Maternal Fetal Medicine, Department of Obstetrics and Gynaecology, University of British Columbia; Julie E van Schalkwyk, MD, Study Director — Clinical Assistant Professor, Division of General Gynaecology & Obstetrics, Department of Obstetrics and Gynaecology, University of British Columbia; Michael WH Suen, MD, Study Director — Resident, Department of Obstetrics and Gynaecology, University of British Columbia
Locations (1):
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada